CLINICAL TRIAL: NCT00376909
Title: New York Prevention Care Manager Project
Brief Title: A Telephone-Based Prevention Care Manager in Increasing Screening Rates for Breast Cancer, Cervical Cancer, and Colorectal Cancer in Minority and Low-Income Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDR0000450797; R01CA087776 (NIH); DMS-15524
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2006-09

CONDITIONS: Breast Cancer; Cervical Cancer; Colorectal Cancer
Keywords: breast cancer; cervical cancer; colon cancer; rectal cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Series of telephone support calls from a trained prevention care manager
  Interventions: Other: educational intervention; Other: study of socioeconomic and demographic variables
- Usual Care (No Intervention): Usual care

INTERVENTIONS:
Other: educational intervention
  Arms: Intervention
Other: study of socioeconomic and demographic variables
  Arms: Intervention

SUMMARY:
RATIONALE: Studying the barriers that prevent minority and low-income women from undergoing cancer screening, and offering encouragement to them over the telephone, may help improve cancer screening rates.

PURPOSE: This randomized phase II trial is studying how well a telephone-based Prevention Care Manager increases screening rates for breast cancer, cervical cancer, and colorectal cancer in minority and low-income women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether telephone support for patients, provided through a Prevention Care Manager (PCM), can increase breast, cervical, and colorectal cancer screening rates among minority and low-income women.
* Measure the amount of PCM time required to improve early cancer detection provided to age-eligible ethnically diverse women seen in community health centers in the New York City area.
* Learn barriers faced by this population in obtaining indicated services (mammograms, Pap tests, fecal occult blood testing, and sigmoidoscopy).
* Assess at baseline and follow-up the office environment and work processes in each participating center (in PCM randomized controlled study only).
* Develop and implement the PCM intervention to help patients overcome barriers.
* Evaluate the impact and costs of the PCM in a randomized controlled efficacy trial.

OUTLINE: This is a randomized, controlled, single-blind, multicenter study. Patients are randomized according to participating center.

* Part 1: Some patients undergo a series of structured interviews about the obstacles to early cancer detection. Participating sites are assessed for study eligibility.
* Part 2: Pilot testing, training, and competency testing of the Prevention Care Managers (PCM) are conducted.
* Part 3: Patients are randomized to 1 of 2 intervention arms.

  * Arm I: Patients are offered health education and follow-up services by telephone with a PCM.
  * Arm II: Patients receive usual care.

PROJECTED ACCRUAL: A total of 2,729 (1,413 for PCM randomized controlled study and 1,316 for pilot study) patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients enrolled in the Prevention Care Manager (PCM) controlled, randomized clinical trial (RCT) must meet the following criteria:

  * Registered to receive care at a participating Community Health Center for at least 6 months
  * Overdue for at least one cancer screening as per the following time periods:

    * No mammography within the past 12 months
    * No Pap test within the past 12 months
    * No home fecal occult blood test within the past 12 months
    * No sigmoidoscopy within the past 5 years
    * No colonoscopy within the past 10 years
  * Must not plan to move out of area or change Community Health Center within 15 months
  * No unresolved, urgent abnormal cancer screening result found in medical record
* Patients enrolled in the PCM dissemination pilot study through Affinity Health Plan must meet the following criteria:

  * Enrolled with Affinity Health Plan for at least 12 months
  * Overdue for at least one cancer screening as per the following time periods:

    * No mammography within the past 2 years
    * No Pap test within the past 3 years
    * No home fecal occult blood test within the past year for women ≥ 50 years old
    * No sigmoidoscopy within the past 5 years
    * No colonoscopy within the past 10 years
  * Must have received care at 1 of 6 participating Community Health Centers in New York City

PATIENT CHARACTERISTICS:

* Female
* Must not be in acute distress or have an acute illness
* Age 50 to 69 years for controlled study patients
* Age 40 to 69 years for pilot study patients

PRIOR CONCURRENT THERAPY:

* No concurrent chemotherapy or radiotherapy
* No concurrent active cancer treatment
* No concurrent palliative care

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2729 (Estimated)
Dates: Start 2001-11; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Follow-up patient cancer 3 months after completion of study treatment
Screening rates as measured by mammography, Pap test, hfoBT, sigmoidoscopy, barium enema and colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Allen J. Dietrich, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (2):
- United States (2):
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Clinical Directors Network, Incorporated, New York, New York

REFERENCES:
- [Result] Dietrich AJ, Tobin JN, Cassells A, Robinson CM, Greene MA, Sox CH, Beach ML, DuHamel KN, Younge RG. Telephone care management to improve cancer screening among low-income women: a randomized, controlled trial. Ann Intern Med. 2006 Apr 18;144(8):563-71. doi: 10.7326/0003-4819-144-8-200604180-00006. PMID 16618953
- [Result] Dietrich AJ, Tobin JN, Cassells A, Robinson CM, Reh M, Romero KA, Flood AB, Beach ML. Translation of an efficacious cancer-screening intervention to women enrolled in a Medicaid managed care organization. Ann Fam Med. 2007 Jul-Aug;5(4):320-7. doi: 10.1370/afm.701. PMID 17664498
- [Result] Ogedegbe G, Cassells AN, Robinson CM, DuHamel K, Tobin JN, Sox CH, Dietrich AJ. Perceptions of barriers and facilitators of cancer early detection among low-income minority women in community health centers. J Natl Med Assoc. 2005 Feb;97(2):162-70. PMID 15712779